CLINICAL TRIAL: NCT04249076
Title: A Phase 3, Multicenter, Randomized, Double-Masked Clinical Trial to Assess the Efficacy and Safety of Clobetasol Propionate Ophthalmic Nanoemulsion 0.05% Compared to Placebo in the Treatment of Inflammation and Pain Associated With Cataract Surgery
Brief Title: Clobetasol Propionate Ophthalmic Nanoemulsion 0.05% for the Treatment of Inflammation and Pain Associated With Cataract Surgery (CLOSE-2)
Acronym: CLOSE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLOBOF3-16IA02
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-11

CONDITIONS: Cataract
Keywords: Cataract Surgery; Inflammation; Pain; Clobetasol propionate; Ophthalmology
MeSH Terms: conditions — Cataract; Inflammation; Pain | interventions — Clobetasol

STUDY DESIGN:
Intervention Model Description: At least 210 participants Will be randomized in a 2:1 randomization ratio (140 to clobetasol arm, 70 to placebo arm) in order to have 202 evaluable participants (4% lost to follow-up rate expected)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Clobetasol propionate (Experimental): First dose of the drug will be dispensed at the end of the Baseline visit at the study center. Then, study medication will be dispensed to the participant for self-administration at a dosage ofe one drop four (4) times a day during 14 days
  Interventions: Drug: Clobetasol Propionate
- Vehicle (Placebo Comparator): First dose of the drug will be dispensed at the end of the Baseline visit at the study center. Then, study medication will be dispensed to the participant for self-administration at a dosage ofe one drop four (4) times a day during 14 days
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Clobetasol Propionate — Clobetasol propionate ophthalmic nanoemulsion 0.05% is an oil-in-water (o/w), clear or slightly yellowish nanoemulsion containing the active ingredient clobetasol propionate at a concentration of 0.05% weight per weight (w/w)
  Other Names: Clobetasol propionate ophthalmic nanoemulsion 0.05%; SVT-15473
  Arms: Clobetasol propionate
Drug: Vehicle — Vehicle is identical in appearance and composition to clobetasol propionate ophthalmic nanoemulsion 0.05% but, without the active substance
  Arms: Vehicle

SUMMARY:
Cataract surgery is one of the most common surgical procedures performed worldwide. In fact, in 2017, 3.8 million cataracts procedures were performed in the US.

Despite of surgical advances, pain and inflammation after ophthalmic surgery continues to be a burden on both patients and physicians. The treatment of postoperative pain is essential for hospitalized patients, but it is even more important for patients who are treated on an outpatient basis.

This study will compare the efficacy and safety of clobetasol propionate ophthalmic nanoemulsion 0.05% to placebo, when administering one drop four times a day during 14 days after routine unilateral cataract surgery. Participants will undergo routine cataract surgery according to the ophthalmologist's normal procedures.

Overall, 210 participants are planned to take part in the study. They will be screened across 20 centers in the US. Participants who experience postoperative inflammation on the first day following routine cataract surgery and who meet all other eligibility criteria will be randomly assigned by chance to one of two study groups in a 2:1 ratio to receive either clobetasol propionate ophthalmic nanoemulsion 0.05 % (N=140) or placebo (N=70) for the treatment of inflammation and pain associated with cataract surgery.

Six (6) study visits are planned: Visit -1 (Screening), Visit 1 (Baseline; 24h after the surgery), Visit 2 (Day 3), Visit 3 (Day 8), Visit 4 (Day 15), and Visit 5 (Day 29).

The ophthalmologist will administer the first dose of the study medication 24 hours after the surgery, at the end of the Baseline visit, at the study center. Study medication will be then dispensed to patients for self-administration during the study at a dosage of one drop four times a day, during 14 days.

Direct instillation is the most efficient method for delivery to the ocular surface and is an accepted and widely used method for topical application to the eye. This study will examine effect and tolerability for 14 days of clobetasol propionate ophthalmic nanoemulsion 0.05% dosed four times a day.

This study is being conducted to support an application for approval to market clobetasol propionate ophthalmic nanoemulsion 0.05% in the US for the indication of inflammation and pain after ocular surgery. The reference (comparator) product in this study, the vehicle, is expected to provide a lower efficacy rate when compared to clobetasol 0.05%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older on day of consent
2. Participants with routine unilateral cataract surgery on the day prior to study randomization
3. Participants with at least 5 cells in anterior chamber on the first day after surgery (at Baseline visit)
4. Willing and able to understand and provide written informed consent form (ICF) (at Screening visit)
5. Women who satisfy one of the following:

   1. Are of child-bearing potential who are not pregnant or lactating and who are either abstinent or sexually active on an acceptable method of birth control (methods that can achieve a failure rate of less than 1% per year when used consistently and correctly, like hormonal contraception (oral pills, implantable device, or skin patch), intrauterine device, bilateral tubal occlusion, or double barrier) for at least 4 weeks prior to Baseline visit and throughout the study (i.e., until Day 29),

OR

Are post-menopausal (have had no menstrual cycle for at least one year prior to Screening visit) or have undergone a sterilization procedure (bilateral tubal ligation, hysterectomy, hysterectomy with unilateral or bilateral oophorectomy or bilateral oophorectomy) at least 6 months prior to Screening visit

Exclusion Criteria:

1. Systemic administration of any corticosteroid or immunosuppressant drugs in the previous 2 weeks prior to the first instillation of the investigational medical product (IMP)
2. Periocular injection in the study eye of any corticosteroid solution within 4 weeks prior to the first instillation of the IMP, or of any corticosteroid depot within 2 months prior to the first instillation of the IMP (Ozurdex® [dexamethasone]: within prior 6 months; Iluvien® [fluocinolone]: within prior 36 months)
3. Instillation of any topical ocular corticosteroid, non-steroidal antiinflammatory drug (NSAID), mast cells stabilizers, antihistamines or decongestants within 2 weeks prior to the first instillation of the IMP, except pre-surgical and/or surgical administration of 1 drop of a topical NSAID or corticosteroid, at the investigator discretion
4. Prescription of any topical ocular medication, except preservative-free antibiotics for prophylactic purposes
5. Any history of glaucoma or ocular hypertension in the study eye
6. History or presence of endogenous uveitis
7. Any current corneal abrasion or ulceration
8. Any confirmed or suspected active viral, bacterial, or fungal keratoconjunctival disease
9. Known hypersensitivity or contraindication to the study drug or any of its components
10. History of steroid-related intraocular pressure (IOP) increase
11. Previous surgery in the last 4 weeks prior to the Screening visit or new surgery scheduled to be performed before the end of the study period on the contralateral eye
12. Presence of ocular hemorrhage which interferes with the evaluation of post-surgery inflammation
13. Presence of intraoperative complications during the cataract surgical procedure that may increase post-operative inflammation; this includes, in particular, patients with ocular hemorrhage, floppy iris syndrome, increased IOP (≥24 mmHg), posterior capsule rupture and injections of gas into the vitreous body
14. Increased cumulative dissipated energy value during phacoemulsification (increased energy used for phacoemulsification exert additional stress on iris and other anterior chamber structures and may generate excessive inflammation)
15. Presence of zonular dialysis (rupture of zonular fibers that attach lens to the ciliar body which may lead to partial luxation of the lens / lens capsule and is a serious complication of cataract surgery)
16. Presence of Fuchs´ endothelial dystrophy (loss of endothelial cells that may result in chronic corneal edema after cataract surgery especially if high energy was used during phacoemulsification)
17. Presence of cornea guttata
18. Pupil dilation lower than 4.5 mm
19. Presence of lower lacrimal duct obstruction and/or history of infectious dacryocystitis
20. Presence of IOP ≥24 mmHg at Baseline visit
21. Participation in any study of an investigational topical or systemic new drug or device within 30 days prior to the Screening visit, or at any time during the study
22. Prior participation in the study described in this protocol, unless patient was not randomized
23. In the opinion of the investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops
24. Disease, condition (including monocular participants), or disorder that in the judgement of investigator could confound study assessments or limit compliance to study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schwartz, MD, Principal Investigator — Director of refractive surgery and laser vision correction at 5th Avenue Eye Associates
Locations (18):
- United States (18):
  - Walman Eye Center, Sun City, Arizona
  - Inland Eye Specialists, Hemet, California
  - United Medical Research Institute, Inglewood, California
  - Visionary Eye Institute, Newport Beach, California
  - North Bay Eye, Petaluma, California
  - Levenson Eye Associates, Jacksonville, Florida
  - International Eye Associates, PA, Ormond Beach, Florida
  - Andrew Gardner Logan dba Ophthalmic Research LLC, Tamarac, Florida
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Ophalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care Ltd, Washington, Missouri
  - NV Eyey Surgery, Henderson, Nevada
  - Houston Eye Associates, Houston, Texas
  - Shah Eye Center, Mission, Texas
  - Braverman-Terry-Oei Eye Associates, San Antonio, Texas
  - Stacy R. Smith, M.D., P.C., Salt Lake City, Utah
  - Virgina Eye Consultants, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coppens M, Versichelen L, Mortier E. Treatment of postoperative pain after ophthalmic surgery. Bull Soc Belge Ophtalmol. 2002;(285):27-32. PMID 12442340
- [Background] Porela-Tiihonen S, Kaarniranta K, Kokki H. Postoperative pain after cataract surgery. J Cataract Refract Surg. 2013 May;39(5):789-98. doi: 10.1016/j.jcrs.2013.03.012. PMID 23608571
- [Background] Patel A, Cholkar K, Agrahari V, Mitra AK. Ocular drug delivery systems: An overview. World J Pharmacol. 2013;2(2):47-64. doi: 10.5497/wjp.v2.i2.47. PMID 25590022
- [Background] Bourlais CL, Acar L, Zia H, Sado PA, Needham T, Leverge R. Ophthalmic drug delivery systems--recent advances. Prog Retin Eye Res. 1998 Jan;17(1):33-58. doi: 10.1016/s1350-9462(97)00002-5. PMID 9537794
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Pascolini D, Mariotti SP. Global estimates of visual impairment: 2010. Br J Ophthalmol. 2012 May;96(5):614-8. doi: 10.1136/bjophthalmol-2011-300539. Epub 2011 Dec 1. PMID 22133988
- [Result] Chiquet C, Aptel F, Creuzot-Garcher C, Berrod JP, Kodjikian L, Massin P, Deloche C, Perino J, Kirwan BA, de Brouwer S, Combette JM, Behar-Cohen F. Postoperative Ocular Inflammation: A Single Subconjunctival Injection of XG-102 Compared to Dexamethasone Drops in a Randomized Trial. Am J Ophthalmol. 2017 Feb;174:76-84. doi: 10.1016/j.ajo.2016.10.012. Epub 2016 Nov 1. PMID 27810317
- [Result] Henzler D, Kramer R, Steinhorst UH, Piepenbrock S, Rossaint R, Kuhlen R. Factors independently associated with increased risk of pain development after ophthalmic surgery. Eur J Anaesthesiol. 2004 Feb;21(2):101-6. doi: 10.1017/s0265021504002042. PMID 14977340
- [Result] Kessel L, Tendal B, Jorgensen KJ, Erngaard D, Flesner P, Andresen JL, Hjortdal J. Post-cataract prevention of inflammation and macular edema by steroid and nonsteroidal anti-inflammatory eye drops: a systematic review. Ophthalmology. 2014 Oct;121(10):1915-24. doi: 10.1016/j.ophtha.2014.04.035. Epub 2014 Jun 14. PMID 24935281
- [Result] Juthani VV, Clearfield E, Chuck RS. Non-steroidal anti-inflammatory drugs versus corticosteroids for controlling inflammation after uncomplicated cataract surgery. Cochrane Database Syst Rev. 2017 Jul 3;7(7):CD010516. doi: 10.1002/14651858.CD010516.pub2. PMID 28670710
- [Result] Sherif Z, Pleyer U. Corticosteroids in ophthalmology: past-present-future. Ophthalmologica. 2002 Sep-Oct;216(5):305-15. doi: 10.1159/000066189. No abstract available. PMID 12424394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with routine unilateral cataract surgery on the day prior to study randomization.
Pre-assignment Details: Patients with at least 5 cells in anterior chamber on the first day after surgery (at Visit 1)
Groups:
- Clobetasol Propionate: Investigational treatment
  1 drop four times a day
- Placebo: Vehicle
  1 drop four times a day
Period: Overall Study
Arm/Group | Clobetasol Propionate | Placebo
Started | 141 | 74
Completed | 139 | 69
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobetasol Propionate | Placebo | Total
Number analyzed (Participants) | 141 | 74 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (8.2) | 67.5 (9.2) | 67.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 45 | 121
  Male | 65 | 29 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 14 | 35
  White | 104 | 52 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Grade
Description: Percentage of participants with anterior chamber cell grade of "0" (absence of cells)
Time Frame: Day 8
Population: FAS Population at Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Clobetasol Propionate | Placebo
Number analyzed (Participants) | 139 | 71
Participants | 38 | 7

2. Secondary Outcome: Pain Visual Analogue Scale (VAS) Score
Description: Percentage of participants with VAS pain score of "0" (no eye pain)
Time Frame: Day 8
Population: FAS Population at Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | Clobetasol Propionate | Placebo
Number analyzed (Participants) | 139 | 71
Participants | 68 | 31

ADVERSE EVENTS:
Time Frame: Overall study period (4 weeks)
Groups:
- Clobetasol Propionate: Interventional treatment
  1 drop four times a day
Arm/Group | Clobetasol Propionate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/141 | 2/74
Other Adverse Events (participants affected / at risk) | 2/141 | 5/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate (N=141) | Placebo (N=74)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cystoid Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate (N=141) | Placebo (N=74)
Corneal oedema (Eye disorders) | 2 (2) | 2 (2)
Eye inflammation (Eye disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication shall be expressly authorized in written by the Sponsor

DOCUMENTS (2):
  • Study Protocol (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT04249076/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04249076/SAP_001.pdf